CLINICAL TRIAL: NCT01881646
Title: Postoperative Neuroinflammation and Cognitive Dysfunction After Abdominal Surgery
Acronym: POPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Lars I Eriksson, Professor, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: POPE
Record Dates: First submitted 2013-06-13; First posted 2013-06-19 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Anesthesia; Surgery; Neurogenic Inflammation; Cognitive Disorders
Keywords: Neuroinflammation; Postoperative cognitive dysfunction
MeSH Terms: conditions — Neurogenic Inflammation; Cognitive Dysfunction; Neuroinflammatory Diseases; Postoperative Cognitive Complications | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positron emission tomography (PET) (Experimental): Positron emission tomography (PET) using [11C]PBR28
  Interventions: Radiation: Positron emission tomography (PET) using [11C]PBR28

INTERVENTIONS:
Radiation: Positron emission tomography (PET) using [11C]PBR28

SUMMARY:
The main purpose of this study is to assess the induction of neuroinflammation in brain regions of interest for learning and memory in adult patients undergoing urological surgery under general anesthesia

DETAILED DESCRIPTION:
The investigators aim to study immune cell activation as a biomarker for neuroinflammation using the cell specific [11C]PBR28 probe as detected by PET imaging techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 60-75 years of age. American Society for Anesthesiologist' criteria (ASA) physical status I-III
2. Lower abdominal surgery (hysterectomy/prostatectomy) under general anaesthesia
3. Obtained consent within 3 months before execution of the study.

Exclusion Criteria:

1. Patient's refusal to participate in the trial
2. Ongoing smoking, snuff or other nicotine compound treatment
3. Disabling neuropsychiatrical disorder (a Mini mental State Examination (MMSE) score ≤ 24, diagnosis of dementia, Mb Alzheimer, Mb Parkinson, schizophrenia, or mental depression) or other signs of significant cognitive decline.
4. History of stroke with neurological sequelae
5. Surgical procedure scheduled for regional anaesthesia.
6. Severe cardia and/or renal and/or hepatic impairment.
7. Coagulopathy.
8. Terminal phase of a chronic disease.
9. Patient on steroidal or non-steroidal anti-inflammatory drugs.
10. Admission B-Glucose > 15 mmol/litre or poorly controlled diabetes mellitus.
11. Presumed uncooperativeness or legal incapacity.
12. Preoperative or later postoperative B-hemoglobin < 90 g/L.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Binding of the PET probe [11C]PBR28 | Preoperatively, once at postoperative day 2-5 and after 3 month
  PET imaging of brain regions of relevance for memory and learning will be compared between the pre- and postoperative states.

SECONDARY OUTCOMES:
Cognitive testing | Preoperatively and after 3 month
  Postoperative cognitive test battery according to the ISPOCD protocol, see Moller JT et al, Lancet 1998.
Inflammatory biomarkers | Preoperatively, once at postoperative day 2-5 and after 3 month, i.e. at the same time as the PET investigation
  Inflammatory biomarkers and genetic analysis of inflammatory biomarkers in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Lars I Eriksson, MD,PhD, Professor, Principal Investigator — Karolinska University Hospital and Karolinska Institutet